CLINICAL TRIAL: NCT01731730
Title: Study to Evaluate the Safety & Efficacy of a Single Intrathecal Pre-Operative Administration of AYX1 Injection at Two Dose Levels Compared to Placebo in Patients Undergoing Unilateral Total Knee Arthroplasty (TKA)
Brief Title: Study to Evaluate Safety/Efficacy of a Single Pre-Op Dose of AYX1 Injection to Treat Pain After Knee Replacement Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adynxx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADYX-002
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Postsurgical Pain
Keywords: Postsurgical pain; Total knee arthroplasty; Total knee replacement
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Vehicle) Injection (Placebo Comparator): Single Intrathecal (spinal) administration of Placebo Injection just prior to intrathecal administration of spinal anesthetic for knee surgery
  Interventions: Drug: Placebo Injection
- AYX1 Injection 110 mg (Experimental): Single Intrathecal (spinal) administration of AYX1 Injection (110 mg) just prior to intrathecal administration of spinal anesthetic for knee surgery
  Interventions: Drug: AYX1 Injection 110 mg
- AYX1 Injection 330 mg (Experimental): Single Intrathecal (spinal) administration of AYX1 Injection (330 mg) just prior to intrathecal administration of spinal anesthetic for knee surgery
  Interventions: Drug: AYX1 Injection 330 mg

INTERVENTIONS:
Drug: Placebo Injection — 3mL solution for intrathecal injection; Vehicle formulation designed to mimic AYX1 Injection (with no active drug)
  Arms: Placebo (Vehicle) Injection
Drug: AYX1 Injection 110 mg — 3mL solution for intrathecal injection with 110 mg of AYX1
  Arms: AYX1 Injection 110 mg
Drug: AYX1 Injection 330 mg — 3mL solution for intrathecal injection with 330 mg of AYX1
  Arms: AYX1 Injection 330 mg

SUMMARY:
The objectives of this proof of concept study are to evaluate the safety and preventive analgesic efficacy of a single preoperative intrathecal administration of AYX1 Injection in patients undergoing unilateral total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo primary unilateral TKA for painful osteoarthritis
* American Society of Anesthesiologists Physical Status Classification System ≤ 3
* Medically stable as determined by the Investigator based on pre-study medical history, physical/neurological examination, clinical lab tests, and 12-lead ECG findings
* Body mass index of 18-40 kg/m2
* Stable medical regimen for ≥ 1 month before randomization
* Able to read and understand study instructions in English, and willing and able to comply with all study procedures

Exclusion Criteria:

* More than 2 other current focal areas of pain, none greater in intensity than the target knee and no other active chronic pain conditions that would compromise operative knee pain evaluation
* Inflammatory arthridities (i.e., rheumatoid arthritis, lupus, ankylosing spondylitis, psoriatic arthritis, gout)
* Operative arthroscopy in the surgical knee in the last 6 months, or other prior surgery in either knee in the last 12 months, except for diagnostic arthroscopy
* Planned use of any of the following for TKA: general endotracheal anesthesia (GETA), peripheral nerve block (i.e., femoral nerve block), neuroaxial (intrathecal or epidural) opioids postoperatively, or knee capsule injections
* Received aspirin within 1 week of randomization, or any nonsteroidal anti-inflammatory drug (NSAID) within 5 half-lives prior to randomization, or planned use of NSAIDS post-operatively through Day 28
* Use of more than 20 mg per day (on average) of oral morphine or its equivalent within 1 month prior to randomization
* Use of adjuvant analgesics for chronic pain control (i.e., gabapentin, pregabalin) during the month prior to randomization or planned use post-operatively through Day 28
* Daily use of benzodiazepines in the 3 months prior to randomization (unless used for sleep and dosage will be consistent after surgery)
* Use of systemic corticosteroids (does not include inhaled steroids) within 3 months or intra-articular steroid injections within 1 month prior to randomization, or planned use of either post-op through Day 28
* Treatment with antibiotics or antivirals (EXCEPTION: topical treatments), immunosuppressives, antipsychotics, anticholinergics, or anticonvulsants within 1 month of randomization, with the exception of prescribed pre-surgical prophylactic antibiotics, and aspirin for cardiac prophylaxis (as long as discontinued within 1 week of randomization
* Current neurologic disorder, which could confound the assessment of pain (i.e., Parkinson's, Multiple Sclerosis)
* Current active depression symptoms
* Has had a change in dose or regimen of SSRIs or SNRIs for depression within 1 month of randomization
* Mini Mental State Exam score < 24 at screening
* Current history of insulin dependent diabetes mellitus, or autoimmune conditions
* Severe chronic obstructive or restrictive pulmonary disease, current diagnosis of obstructive sleep apnea documented by a sleep laboratory study, or current home use of continuous positive airway pressure (CPAP) or bi-level positive airway pressure (BIPAP)
* Current evidence of alcohol abuse or history of alcohol-related complications within 1 year of randomization
* Known or suspected history of illicit drug abuse within 1 year before randomization, current or planned use of medical marijuana, or history of opioid dependence within 2 years before randomization
* Any malignancy within the past year, with the exception of basal cell carcinoma or uncomplicated or stable skin cancers documented to not require further or immediate treatment
* Women who are pregnant or nursing

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pain with walking during 5 meter walk test | 0-48 hours after surgery
  Mean pain rating on the Numerical Rating Scale (NRS) with walking during the 5 meter walk test during inpatient stay 0-48 hours
Pain with walking during 15 meter walk test | From hospital discharge to Day 28
  Mean pain rating on the Numerical Rating Scale (NRS) with walking during the 15 meter walk test during outpatient period up to Day 28

SECONDARY OUTCOMES:
Total use of opioid medications (morphine equivalents) during hospital stay | 0-48 hours after surgery
Total use of opioid medications (morphine equivalents) post-discharge to Day 28 | From hospital discharge to Day 28
Pain with 45 degrees of knee flexion | 0-48 hours after surgery
  Mean pain rating on the Numerical Rating Scale (NRS) for 45 degrees active knee flexion
Pain with 90 degrees of knee flexion | From 7 to 28 days after surgery
  Mean pain rating on the Numerical Rating Scale (NRS) for 90 degrees active knee flexion

OTHER OUTCOMES:
Brief Pain Inventory functional interference scores at Days 7, 14, 21, 28, and 42 | 7 to 42 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Donald C Manning, MD, PhD, Study Director — Adynxx, Inc.
Locations (7):
- United States (7):
  - Sheffield, Alabama
  - Phoenix, Arizona
  - Boynton Beach, Florida
  - Altoona, Pennsylvania
  - Houston, Texas
  - Nassau Bay, Texas
  - Odessa, Texas